CLINICAL TRIAL: NCT04051788
Title: Effects of 6 Weeks of Step Aerobics Training on Pulmonary Functions Among Females With Sedentary Life Style.
Brief Title: 6 Weeks Step Aerobics Training Among Females With Sedentary Life Style.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RiphahIU Syeda Rida Fatima
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Sedentary Lifestyle
Keywords: Sedentary Lifestyle; Step Aerobics; Pulmonary Function
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step Aerobics (Experimental): Step Aerobics Training (120 to 126 foot steps per min)
  Interventions: Other: Step Aerobics
- Aerobic exercise (Lower limb Cycling) (Active Comparator): Lower Limb Aerobic cycling
  Interventions: Other: Aerobic exercise (Lower limb Cycling)

INTERVENTIONS:
Other: Step Aerobics — Alternating step knee-lift sequences; alternating leg up, up, down, down patterns; and step kicks, 120 to 126 foot strikes per minute, 20 to 30 minutes per session s, 3 sessions per week up to 6 weeks,The target intensity for all sessions will set at 50-70% heart rate (HR) reserve.
  Arms: Step Aerobics
Other: Aerobic exercise (Lower limb Cycling) — Lower Limb Aerobic cycling, 20 to 30 minutes per session, 3 sessions per week up to 6 weeks, The target intensity for all sessions will set at 50-70% heart rate (HR) reserve
  Arms: Aerobic exercise (Lower limb Cycling)

SUMMARY:
To determine the Effects of 6 weeks of Step Aerobics Training on Pulmonary Functions among females with sedentary life style. Traditional aerobic training programs has great effects to improved pulmonary functions in individuals with sedentary life style but on the other hand there is another type of aerobic training named step aerobic which is different from traditional training up-to knowledge has less work on pulmonary function but effective on functional score, and walking velocity this gap further need to identify. This study will help us to choose either of training program to get maximum beneficial outcomes particularly on pulmonary function test on female students with sedentary life style.

DETAILED DESCRIPTION:
A sedentary lifestyle is defined as an individual living with very little or no physical activity. In daily routine the person spending most of his or her time in watching television, playing games on mobile ,using internet, reading books , often sitting or lying down while doing these activities. It can lead to many health problems and potentially very harmful.

Aerobic exercise is defined as physical exertion that depends upon energy generating process. Aerobic defined as something relating to and involving which required free oxygen. During aerobic exercise maximum use of oxygen can meet the energy demand of the body.

Activities with light to moderate intensities that adequately meet the demands of aerobic metabolism, this can be performed for long period of times.There is a term use aerobic exercise that is "solely" aerobic which is defined as low intensity is required to consumed all carbohydrates in the body and termed them into energy. According to this ,some common examples of aerobic exercise that are walking , swimming , jogging, running and cycling.

Aerobic has great impact on decrease the severity of depression and anxiety . Another study on people who are suffered from depression , asked them to walk for 30 minutes on treadmill and reassess them after 10 days. The results shows significant increase and improvement in their mood and reduction in overall depression episodes and symptoms, they feel fresh and more alive start participate in daily activities . Their negative thoughts which make them depressive also get reduced to some extent .The results shows that physical activity or exercise only for a short period of time may give you a boost in your mood and overall health status. Only a single exercise session has a great impact on the overall mental health.

Another research was conducted on target matching foot stepping to evaluate the proprioception and function of knee osteoarthritis . It includes functional score , walking velocity and overall knee performance to determine the efficacy of knee osteoarthritis. The exercise was designed to perform in sitting position as knee arthritic patients are not able to tolerate in standing position.

ELIGIBILITY:
Inclusion Criteria:

* Female students
* Sedentary life style (low Physical activity)

Exclusion Criteria:

* Asthmatic patients
* Any history of Malignancies.
* Students with psychiatric disorders
* Musculoskeletal disease that he was unable to perform aerobic exercises
* Neuromuscular diseases that patient was unable to maintain balance

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — That was because of female sedentary nature in Pakistan which has our objective to meet.
Enrollment: 80 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 6th week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 6th week
  Changes From the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters.
Peak Expiratory Flow (PEF) | 6th Week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.

SECONDARY OUTCOMES:
Oxygen Saturation (SpO2) | 6th week
  Changes from baseline SPO2 was measured in percentage. Oxygen immersion is the division of oxygen-soaked hemoglobin with respect to add up to hemoglobin in the blood. Pulse oximeter measure it.
Pulse Rate | 6th week
  Changes from baseline, Pulse rate was measured per minute through pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilmore JH. Aerobic exercise and endurance: improving fitness for health benefits. Phys Sportsmed. 2003 May;31(5):45-51. doi: 10.3810/psm.2003.05.367. PMID 20086470
- [Background] Hallage T, Krause MP, Haile L, Miculis CP, Nagle EF, Reis RS, Da Silva SG. The effects of 12 weeks of step aerobics training on functional fitness of elderly women. J Strength Cond Res. 2010 Aug;24(8):2261-6. doi: 10.1519/JSC.0b013e3181ddacc6. PMID 20634751
- [Background] Jan MH, Tang PF, Lin JJ, Tseng SC, Lin YF, Lin DH. Efficacy of a target-matching foot-stepping exercise on proprioception and function in patients with knee osteoarthritis. J Orthop Sports Phys Ther. 2008 Jan;38(1):19-25. doi: 10.2519/jospt.2008.2512. PMID 18357655
- [Background] Khaled M B, A M, S T K, S P C, R D. Effect of traditional aerobic exercises versus sprint interval training on pulmonary function tests in young sedentary males: a randomised controlled trial. J Clin Diagn Res. 2013 Sep;7(9):1890-3. doi: 10.7860/JCDR/2013/5797.3343. Epub 2013 Sep 10. PMID 24179890
- [Background] Moradians V, Rahimi A, Javad Moosavi SA, Sahebkar Khorasani FS, Mazaherinejad A, Mortezazade M, Raji H. Effect of Eight-Week Aerobic, Resistive, and Interval Exercise Routines on Respiratory Parameters in Non-Athlete Women. Tanaffos. 2016;15(2):96-100. PMID 27904541
- [Background] Cheng YJ, Macera CA, Addy CL, Sy FS, Wieland D, Blair SN. Effects of physical activity on exercise tests and respiratory function. Br J Sports Med. 2003 Dec;37(6):521-8. doi: 10.1136/bjsm.37.6.521. PMID 14665592
- [Background] Larson JL, Covey MK, Wirtz SE, Berry JK, Alex CG, Langbein WE, Edwards L. Cycle ergometer and inspiratory muscle training in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1999 Aug;160(2):500-7. doi: 10.1164/ajrccm.160.2.9804067. PMID 10430720
- [Background] Garrod R, Dallimore K, Cook J, Davies V, Quade K. An evaluation of the acute impact of pursed lips breathing on walking distance in nonspontaneous pursed lips breathing chronic obstructive pulmonary disease patients. Chron Respir Dis. 2005;2(2):67-72. doi: 10.1191/1479972305cd068oa. PMID 16279153
- [Background] Spahija J, de Marchie M, Grassino A. Effects of imposed pursed-lips breathing on respiratory mechanics and dyspnea at rest and during exercise in COPD. Chest. 2005 Aug;128(2):640-50. doi: 10.1378/chest.128.2.640. PMID 16100149